CLINICAL TRIAL: NCT05193786
Title: Low Versus High PEEP in Noninvasive Ventilation for Hypoxemic Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Duan jun, Principal Investigator, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChongqingMU5
Record Dates: First submitted 2021-12-20; First posted 2022-01-18 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Low versus high PEEP
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low PEEP group (Active Comparator): In low PEEP group, the PEEP was 5 cmH2O and inspiratory pressure was 10-20 cmH2O in noninvasive ventilation.
  Interventions: Procedure: Different level of PEEP
- High PEEP group (Experimental): In high PEEP group, the PEEP was 10-15 cmH2O and inspiratory pressure was 15-20 cmH2O in noninvasive ventilation.
  Interventions: Procedure: Different level of PEEP

INTERVENTIONS:
Procedure: Different level of PEEP — Different level of PEEP (low versus high) was applied in noninvasive ventilation.

SUMMARY:
Current study aimed to explore the effect of high PEEP during noninvasive ventilation among hypoxemic patients with acute respiratory failure.

DETAILED DESCRIPTION:
This was a 1:1 randomized control trial to explore the effect of high versus low PEEP in noninvasive ventilation hypoxemic patients with acute respiratory failure. Several ICUs in China performed this study. In the high PEEP group, the PEEP maintained at 10-15 cmH2O, the inspiratory pressure maintained at 15-20 cmH2O. In the low PEEP group, the PEEP maintained at 5 cmH2O, the inspiratory pressure maintained at 10-20 cmH2O. The primary outcome was incidence of noninvasive ventilation failrue.

ELIGIBILITY:
Inclusion Criteria

* age between 16 and 85 years
* use of dedicated noninvasive ventilator
* PaCO2 ≤50 mmHg
* PaO2/FiO2 ≤300mmHg
* expectation of noninvasive ventilation >12 hours
* consciousness (Kelly score ≤3 or GCS≥13)

Exclusion Criteria

* use of noninvasive ventilation before randomization > 24 hours
* use of noninvasive ventilation due to heart failure, asthma, acute excerbation of COPD
* presence of contraindication of noninvasive ventilation such as malformation, rencent pulmonary or esophageal surgery et al.
* end stage disease (expectation of life < 6 months)
* pneumothorax
* noninvasive ventilation intolerance
* refusal of paticipation
* pregant woman
* requirement of emergency intubation

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of noninvasive ventilation failure | From randomization to 28 days of study
  Noninvasive ventilation failure was defined as intubation, death or withdrawal of therapy during noninvasive ventilation.

SECONDARY OUTCOMES:
28-day mortality | From randomization to 28 days of study
  Died within 28 days of study
Duration of noninvasive ventilation | From beginning to 28 days of study
  The days spent on noninvasive ventilation
Duration of invasive mechanical ventilation | From randomization to 28 days of study
  The days spent on invasive ventilation
Length of stay in ICU | From beginning to 28 days of study
  The days spent in ICU
Length of stay in hospital | From beginning to 28 days of study
  The days spent in hospital
The changes of PaO2/FiO2 | From randomization to 28 days of study
  Oxygenation was calculated as PaO2/FiO2.
Side effect | From randomization to 28 days of study
  Side effect included the incidence of pressure ulcer, pneumothorax, vomitting, aspiration and dryness

CONTACTS AND LOCATIONS:
Overall Officials: Jun Duan, Dr., Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No